CLINICAL TRIAL: NCT00006371
Title: A Phase II Trial of Early Medical Adrenalectomy for "D0.5" Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12219; NCI-G00-1863 (Other: NCI)
Record Dates: First submitted 2000-10-04; First posted 2004-04-02 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aminoglutethimide; Ketoconazole; Hydrocortisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone with Ketoconazole (Active Comparator): Patients are stratified according to prior antiandrogen therapy (yes vs no). Patients with prior antiandrogen therapy begin study therapy after appropriate antiandrogen withdrawal, while those without such prior therapy begin study therapy immediately. Patients undergo medical adrenalectomy using hydrocortisone combined with ketoconazole. Oral hydrocortisone is administered twice daily. Oral aminoglutethimide is administered twice daily for 1 week and then 4 times daily during subsequent weeks. Oral ketoconazole is administered three times daily.
  Interventions: Drug: ketoconazole; Drug: therapeutic hydrocortisone
- Hydrocortisone with Aminoglutethimide (Active Comparator): Patients are stratified according to prior antiandrogen therapy (yes vs no). Patients with prior antiandrogen therapy begin study therapy after appropriate antiandrogen withdrawal, while those without such prior therapy begin study therapy immediately. Patients undergo medical adrenalectomy using hydrocortisone combined with aminoglutethimide. Oral hydrocortisone is administered twice daily. Oral aminoglutethimide is administered twice daily for 1 week and then 4 times daily during subsequent weeks. Oral ketoconazole is administered three times daily.
  Interventions: Drug: aminoglutethimide; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Drug: aminoglutethimide
  Other Names: Cytadren
  Arms: Hydrocortisone with Aminoglutethimide
Drug: ketoconazole
  Other Names: Nizoral
  Arms: Hydrocortisone with Ketoconazole
Drug: therapeutic hydrocortisone
  Other Names: corticosteroid

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as aminoglutethimide or ketoconazole may stop the adrenal glands from producing hormones. Combining hydrocortisone with either aminoglutethimide or ketoconazole may be an effective treatment for prostate cancer.

PURPOSE: Phase II trial to study the effectiveness of combining hydrocortisone with either aminoglutethimide or ketoconazole in treating patients who have localized stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the Prostate-Specific Antigen (PSA) response proportion and duration of response of patients with localized stage IV (D0.5) adenocarcinoma of the prostate treated with early medical adrenalectomy using hydrocortisone combined with aminoglutethimide or ketoconazole after prior antiandrogen withdrawal. II. Compare the incidence of grades 3-4 toxicities of these regimens in these patients. III. Correlate adrenal androgen suppression with response in these patients.

OUTLINE: Patients are stratified according to prior antiandrogen therapy (yes vs no). Patients with prior antiandrogen therapy begin study therapy after appropriate antiandrogen withdrawal, while those without such prior therapy begin study therapy immediately. Patients undergo medical adrenalectomy using hydrocortisone combined with aminoglutethimide OR ketoconazole. Oral hydrocortisone is administered twice daily. Oral aminoglutethimide is administered twice daily for 1 week and then 4 times daily during subsequent weeks. Oral ketoconazole is administered three times daily. Combination treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the prostate Stage IV (D0.5; no evidence of disease on CT or bone scan after testicular androgen ablation) PSA progression after testicular androgen ablation with or without antiandrogen therapy Progression is defined as at least 2 consecutive rising PSA levels (drawn at least 2 weeks apart) with a greater than 50% rise above the last nadir level (arbitrary PSA at least 2 ng/dL)

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other medical conditions that would increase risk Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: See Disease Characteristics Greater than 4 weeks since prior flutamide (6 weeks for bicalutamide or nilutamide) No prior aminoglutethimide or ketoconazole for prostate cancer Continuation of primary testicular androgen suppression (i.e., LHRH analog) required Radiotherapy: Not specified Surgery: Not specified Other: No concurrent terfenadine, astemizole, cisapride, or other medicines known to interact with ketoconazole

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2000-05; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) for Treatment Arm | 1 year
  Determine the PSA response proportion and duration of response of patients with localized stage IV (D0.5) adenocarcinoma of the prostate treated with early medical adrenalectomy using hydrocortisone combined with aminoglutethimide or ketoconazole after prior antiandrogen withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Fishman, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States